CLINICAL TRIAL: NCT03142165
Title: A Randomized, Placebo-Controlled, Double-Blind, Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BMS-986263 in Healthy Participants
Brief Title: A Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BMS-986263 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: IM025-001
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Fibrosis
MeSH Terms: conditions — Fibrosis | interventions — Diphenhydramine; Famotidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BMS-986263 (Experimental)
  Interventions: Drug: BMS-986263; Drug: Diphenhydramine; Drug: Famotidine
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo; Drug: Diphenhydramine; Drug: Famotidine

INTERVENTIONS:
Drug: BMS-986263 — 3 weekly doses of 90 mg infused intravenous administration
  Arms: BMS-986263
Other: Placebo — Placebo
  Arms: Placebo
Drug: Diphenhydramine — 50 mg intravenous administration
Drug: Famotidine — 20 mg intravenous administration

SUMMARY:
The purpose of this study is to assess the safety and tolerability of BMS-986263 in healthy volunteers.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy participants as determined by no clinically significant deviation from normal in medical history, physical exam, ECGs, and clinical laboratory determinations
* Weight within the range of ≥60 and ≤90 kg
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug
* WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with BMS-986263 (21 days), plus 5 half-lives of BMS-986263 (7.5 days) plus 30 days (duration of ovulatory cycle) for a total of 90 days post-treatment completion
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with BMS-986263 (21 days) plus 5 half-lives of BMS-986263 (7.5 days) plus the duration of sperm turnover (90 days) for a total of 118.5 days post-treatment completion. In addition, male participants must be willing to refrain from sperm donation during this time. Azoospermic males are exempt from contraceptive requirements

Exclusion Criteria:

* History or evidence of active infection and/or febrile illness within 7 days of Study Day 1 (e.g., bronchopulmonary, urinary, gastrointestinal, etc.)
* History of serious bacterial, fungal, or viral infections that let to hospitalization and IV antibiotic treatment within 90 days prior to screening, or any recent serious infection requiring antibiotic treatment within 30 days of Study Day 1
* History of recurrent or chronic sinusitis, bronchitis, pneumonia, urinary tract infection, or skin infection (recurrent or chronic infection is defined as ≥2 episodes within a 6 month period)
* Active herpes infection, including herpes simplex 1 and 2 and herpes zoster (demonstrated on physical examination and/or medical history)
* History of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* Presence of active tuberculosis (TB), latent TB, or inadequately treated latent or active TB

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AE) | 28 days
  measured by incidences
Serious Adverse Events (SAE) | 30 days
  measured by incidences
Infusion related reactions | 28 days
  measured by incidences
Abnormalities in clinical laboratory tests | 28 days
  measured by incidences
Abnormal vital sign measurements | 28 days
  measured by incidences
Abnormal electrocardiogram measurements | 28 days
  measured by incidences
Physical examination abnormalities | 28 days
  measured by incidences

SECONDARY OUTCOMES:
Cmax | 28 days
  Maximum observed plasma concentration
Tmax | 28 days
  Time of maximum observed plasma concentration
AUC(0-T) | 28 days
  Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration
AUC(TAU) | 28 days
  Area under the concentration-time curve in one dosing interval (multiple dose only)
T-HALF | 28 days
  Terminal phase half-life
CLT | 28 days
  Total body clearance after IV dose
AI_AUC | 28 days
  Accumulation Index, the ratio of AUC(TAU) at steady-state to that after the first dose (Day 15 only)
T-HALFeff_AUC | 28 days
  Effective elimination half-life that explains the degree of accumulation observed for AUC(TAU) (Day 15 only)
Ctrough | 28 days
  Trough observed plasma concentration
Comparison of pharmacokinetic (PK) parameters in non-Japanese versus Japanese patients | 28 days
  Investigation of population specific differences in PK

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Wcct Global, Llc, Cypress, California, United States

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx